CLINICAL TRIAL: NCT01579695
Title: A Phase 4, Observational, Multicenter, 10-year Prospective Cohort Safety Study Comparing Subjects With HIV-associated Abdominal Lipohypertrophy Exposed to EGRIFTA® (Tesamorelin for Injection) to a Similar Group of Subjects Not Exposed to EGRIFTA®
Brief Title: Long-term Observational Study in HIV Subjects Exposed to EGRIFTA®
Status: Terminated | Type: Observational
Sponsor: Theratechnologies (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR200147-501
Record Dates: First submitted 2012-04-12; First posted 2012-04-18 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: HIV
Keywords: HIV with lipohypertrophy
MeSH Terms: interventions — tesamorelin; Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Exposed Group will receive Tesamorelin
  Interventions: Drug: Tesamorelin for injection
- Control Group will not receive Tesamorelin

INTERVENTIONS:
Drug: Tesamorelin for injection — Daily 2 mg subcutaneous injections of Tesamorelin
  Groups: Exposed Group will receive Tesamorelin

SUMMARY:
The purpose of this observational, 10-year, prospective cohort study is to assess the potential safety concerns of long-term exposure to EGRIFTA® in HIV-infected subjects with abdominal lipohypertrophy compared with a similar group of subjects not exposed to EGRIFTA®.

ELIGIBILITY:
Inclusion Criteria:

All of the following inclusion criteria must be fulfilled:

1. Subject has given written informed consent;
2. Subject is an adult man or woman ≥ 18 years old;
3. Subject has HIV infection;
4. Subject has physical evidence of excess abdominal fat, as determined by the examining study physician.
5. Subject has completed standard of care assessments (mammography, cervical PAP smear, colonoscopy and blood work for HIV-1 RNA, CD4 cell count, renal, hepatic, and hematology, PSA test, fasting blood glucose, lipid panel ) prior to being enrolled onto the study.

Exclusion Criteria:

Exclusion criteria 1 through 4 are based on the contraindications for EGRIFTA®.

1. Disruption of the hypothalamic-pituitary axis, including conditions such as hypophysectomy, hypopituitarism, pituitary tumor/surgery, head irradiation, or head trauma;
2. Active malignancy (newly diagnosed or recurrent)
3. Known hypersensitivity to tesamorelin and/or mannitol
4. Pregnancy or lactation
5. Use of EGRIFTA® within 6 months prior to baseline
6. Failure to complete any standard of care assessments listed in Section 5.2.1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be representative of the HIV-injected population affected by abdominal lipohypertrophy
Sampling Method: Probability Sample
Enrollment: 391 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Time to development of malignancies in HIV-infected subjects with abdominal lipohypertrophy exposed to EGRIFTA® vs. concurrent, comparable control group not exposed to EGRIFTA® | 10 years

SECONDARY OUTCOMES:
Time to development or worsening of Type 2 Diabetes Mellitus, diabetic retinopathy, hypersensitivity reactions, hepatic and renal function, adverse events and major adverse cardiovascular events | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Mamputu, PhD — Theratechnologies Inc.
Locations (30):
- United States (30):
  - Franco Felizarta, MD, Bakersfield, California
  - Pacific Coast Medical Group, Fountain Valley, California
  - University of California CARE Clinic, Los Angeles, Los Angeles, California
  - Tower Infectious Diseases Medical Associates, Los Angeles, California
  - Oasis Clinic, Los Angeles, California
  - VAMC, Infectious Disease Section 111W, San Francisco, California
  - Dupont Circle Physician's Group, Washington D.C., District of Columbia
  - Capital Medical Associates, PC, Washington D.C., District of Columbia
  - Gary J. Richmond, M.D., PA, Fort Lauderdale, Florida
  - The Kinder Medical Group-AHF, Miami, Florida
  - Orange County Health Department, Orlando, Florida
  - Rowan Tree Medical, P.A., Wilton Manors, Florida
  - Absolute Care Medical Center, Atlanta, Georgia
  - Northstar Medical Center, Chicago, Illinois
  - Southern Illnois University School of Medicine, Springfield, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Researth Institute, Springfield, Massachusetts
  - Be Well Medical Center, P.C, Berkley, Michigan
  - Southhampton Clinical Research, Inc. d.b.a. Central West Clinical Research, St Louis, Missouri
  - Southampton Healthcare, Inc., St Louis, Missouri
  - South Jersey Unfectious Disease, Somers Point, New Jersey
  - University at Buffalo, State University of NY, Erie County Medical Center, Buffalo, New York
  - Ricky K. Hsu, MD, PC, New York, New York
  - Summa Health Care System, Akron, Ohio
  - Virginia Mason Medical Center, Tulsa, Oklahoma
  - Reading Hospital and Medical Center, West Reading, Pennsylvania
  - St. Hope Foundation, Inc., Bellaire, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Virginia Mason Medical Center, Seattle, Washington